CLINICAL TRIAL: NCT07408102
Title: Online Study on the Impact of a Self-Help Tool for Social Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Princeton University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18016
Record Dates: First submitted 2025-12-12; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Social Anxiety
Keywords: Cognitive Restructuring; Exposure Therapy; Cognitive Behavioral Therapy; Internet-Based Intervention; Social Anxiety; Predictive Models; Patient-Specific Modeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): All participants are assigned to the e-couch social anxiety program. Over a 5-week study period, participants are instructed to complete specific modules on a weekly schedule. They are asked to engage with the program at least once per week for approximately 30 minutes. Participants receive weekly reminders and guidance indicating which modules to complete each week.
  Interventions: Behavioral: Internet-delivered self-help for social anxiety based on principles of cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Internet-delivered self-help for social anxiety based on principles of cognitive behavioral therapy — Participants will be offered the use of a self-help tool, e-couch (https://ecouch.com.au), for 5 weeks. e-couch is an online, self-directed tool that provides interactive self-help and evidence-based information to help users understand and manage common mental health challenges including symptoms of depression and anxiety. The e-couch social anxiety program will be used in this study. It is structured like an interactive self-help book and participants can log back into at any time to learn and review skills. The e-couch social anxiety program includes a comprehensive information module, as well as self-help modules with interactive exercises and workbooks that teach evidence-based strategies. The content will cover topics such as cognitive restructuring and exposure, with an emphasis on learning strategies to reduce social anxiety.

SUMMARY:
The goal of this clinical trial is to understand which individuals benefit most from an internet-based cognitive behavioral intervention for social anxiety. Adults aged 18-65 will complete a self-guided online program designed to reduce anxiety symptoms. The investigators will use a combination of self-reported clinical information and data from computerized decision-making and cognitive tasks to predict changes in symptom scores from the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Live in the United States
* Comfortable reading and writing in English
* Have regular access to the internet and a desktop/laptop computer
* Report wanting to feel more comfortable in social situations, to improve social confidence, and/or to reduce symptoms of social anxiety as primary reason for joining the study
* Have a valid photo ID and be willing to complete a video-based identity verification call if requested

Exclusion Criteria:

* Lack of attention when completing parts of the study, and/or not completing the study tasks as instructed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Predictive accuracy of change in social anxiety symptom severity, as measured by Liebowitz Social Anxiety Scale (LSAS) total score, from baseline to end of intervention (5 weeks) | Baseline (pre-intervention) to end of intervention (5 weeks)
  Social anxiety symptom severity will be assessed using the Liebowitz Social Anxiety Scale (LSAS), a validated self-report questionnaire measuring fear and avoidance across social interaction and performance situations. The LSAS total score ranges from 0 to 144, with higher scores indicating greater social anxiety symptom severity.
  LSAS total scores will be collected at baseline (pre-intervention) and at the end of the 5-week e-couch intervention period. The outcome metric is the individual-level change in LSAS total score, calculated as the end-of-intervention score minus the baseline score.
  The primary outcome is the accuracy with which pre-intervention self-report measures and computerized behavioral task performance predict change in LSAS total score. Analyses will examine the extent to which individual differences in decision-making and cognitive task performance account for variability in symptom change across participants.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Niv, PhD, Principal Investigator — Princeton University; Jamie C Chiu, PsyD, Principal Investigator — Princeton University
Locations (1):
- Princeton University, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will share de-identified individual participant data used in the results publication, including questionnaire data and data from computerized cognitive and decision-making tasks, with other researchers upon reasonable request and after publication.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Within one year after study completion
Access Criteria: Upon reasonable request and providing that the requesters will treat the data in line with the researchers' ethical principles. Researchers may also make de-identified data publicly available.